CLINICAL TRIAL: NCT06309420
Title: Prospective, Single-blinded, Randomized Trial to Evaluate the Efficacy of a Cryogenic Medical Device in Treatment of Common and Plantar Warts Versus a Comparator Product.
Brief Title: Clinical Trial to Evaluate Efficacy and Safety of a Cryogenic Medical Device for Treatment of Common and Plantar Warts
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oystershell NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19E0566
Record Dates: First submitted 2022-12-16; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Intervention Model Description: Investigator-blinded, Randomized,Tested product versus comparator (benchmark product), In parallel groups, With multiple applications, Single centre.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pixie CO2 (Experimental): Cryogenic treatment of warts (Carbonic ice tablet) Maximum 3 application by the technician in charge of the study Apply 15 seconds for a wart on hand or arm and 40 seconds for a wart on feet or toe
  Interventions: Device: Cryogenic treatment of warts (Pixie CO2)
- Wortie® (Active Comparator): Cryogenic treatment of wart (dimethylether-based product) Maximum 3 application by the technician in charge of the study. Apply 20 seconds for a wart on hand or arm and 40 seconds for a wart on feet or toe
  Interventions: Device: Cryogenic treatment of warts (Wortie®)

INTERVENTIONS:
Device: Cryogenic treatment of warts (Pixie CO2) — Treatment of common and plantar warts by cryotherapy treatment.
  Other Names: X92001686
  Arms: Pixie CO2
Device: Cryogenic treatment of warts (Wortie®) — Treatment of common and plantar warts by cryotherapy treatment.
  Arms: Wortie®

SUMMARY:
The present study was set-up to evaluate clinical efficacy of Pixie CO2 versus a comparator product (Wortie®) for the treatment of common and plantar warts.

DETAILED DESCRIPTION:
The use of cryotherapy has been long known to be effective against warts. The indications for Pixie CO2 are in line with the indications presented in the collected literature data, as well as with the indications of similar devices.

The benefits of the use of cryotherapy for warts is clearly evidenced. The treatment period is short (up to 3 treatments with a 14 day interval, compared to daily application of keratinolytics or fluorouracil, over a period of weeks). The cryotherapy application through a conic applicator is much more precise than with most chemical substances. Chemical substance application is leading to more side effects of the surrounding skin (typical for chemical treatment are pain, blistering, ulceration and contact dermatitis).

The Instructions for Use were developed in line with these data and are therefore covering all hazards known up to the date of this report.

Based on these data the product received its CE-mark approval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject.
* Sex: male or female.
* Age: more than 4 years old.
* Subject presenting at least 1 new common wart on hand or a plantar wart (wart present since less than 6 months) of a size less than 0.8cm.
* Subject, including minors aged more than 16 years, having given freely and expressly his/her informed consent.
* Minor whose legal guardians have given their free and express informed consent.
* Subject who is able to comply with the study requirements, as defined in the present rotocol, at the Investigator's appreciation.
* Subject or child's legal guardians being affiliated to a health social security system.
* Female subject of childbearing potential should use a medically accepted contraceptive regimen (at the Investigator's discretion) since at least 12 weeks before the beginning of the study, during all the study.

Exclusion Criteria:

* Pregnant, parturient, or nursing woman or planning a pregnancy during the study.
* Subject who had been deprived of their freedom by administrative or legal decision.
* Subject in a social or sanitary establishment.
* Major subject who is under guardianship or who is not able to express his consent.
* Subject suspected to be non-compliant according to the Investigator's judgment.
* Subject suffering from a severe or progressive disease or any other pathology that may interfere with the evaluation of the study results.
* Subject with a cutaneous disease other than common and plantar warts, on the studied zone.
* Subject with a known allergy to one of the component of the products or to the comparator.
* Subject who has diabetes.
* Subject having problems with blood circulation, or having a blood clotting condition.
* Subject with immune deficiency or autoimmune disease.
* Subject presenting more than 10 warts on the body.
* Subject presenting bleeding warts.
* Subject presenting birthmarks, moles, warts with hairs growing from them, or any other spots on the treated and surrounding area.
* Subject having a sensitive skin, inflamed, infected, irritated, red, damaged, cut, grazed, diseased or itchy on the treated zone.
* Subject presenting genital warts, flat warts, filiform warts, periungual warts or warts larger than 0.8cm.
* Subject presenting 2 or more warts adjacent to each other.
* Subject undergoing a topical treatment on the test area or a systemic treatment:
* anti-inflammatory medication during the previous 2 weeks and during the study,
* immunosuppressors and/or corticoids during the 4 previous weeks and during the study,
* retinoids during the 6 previous months and during the study,
* any medication stabilized for less than one month.
* Subject who received a treatment of any type on the selected wart during the previous 6 months.
* Intensive exposure to sunlight or UV-rays on the studied zone within the previous month and/or foreseen during the study.
* Subject planning to change her/his life habits during the study.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-11-07 (Actual); Primary Completion 2020-08-10 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Percentage of subjects with clinical wart remission | 1 treatment (Day 0), 2 treatments (Day 15), 3 treatments (Day 30)
  Comparison of the percentage of subjects with clinical wart remission after 1, 2 and 3 treatments with the tested product group versus comparator group, as observed during clinical evaluation of the treated wart by a dermatologist.

SECONDARY OUTCOMES:
Number of treatments | 1 treatment (Day 0), 2 treatments (Day 15), 3 treatments (Day 30)
  Comparison of the number of treatments needed for clinical remission of warts with both products
Efficacy of the freezing process (Surface Area) | Measurement treatment 1 (Day 0), Measurement treatment 2 (Day 15), Measurement treatment 3 (Day 30)
  Surface area measurements of frostbite area to evaluate the efficacy of the freezing process
Diameter of the wart | Before treatment Day 0, after 1 treatment (Day 3 & Day 15), after 2 treatments (Day 30), after 3 treatments (Day 45)
  Macrophotography of the wart
Roughness of the wart | Before treatment Day 0, after 1 treatment (Day 3 & Day 15), after 2 treatments (Day 30), after 3 treatments (Day 45)
  Evaluation of roughness of the wart by blinded dermatologist. Classification scheme was used: 0=absence, 1=light, 2=moderate, 3=severe, and 4=very severe
Thickness of the wart (For common warts only) | Before treatment Day 0, after 1 treatment (Day 3 & Day 15), after 2 treatments (Day 30), after 3 treatments (Day 45)
  Evaluation of thickness of the wart by blinded dermatologist. Classification scheme was used: 0=absence, 1=light, 2=moderate, 3=severe, and 4=very severe
Presence of small dark spot (For plantar warts only) | Before treatment Day 0, after 1 treatment (Day 3 & Day 15), after 2 treatments (Day 30), after 3 treatments (Day 45)
  Evaluation of presence of a small dark spot by blinded dermatologist. Classification scheme was used: 0=absence, 1=light, 2=moderate, 3=severe, and 4=very severe
Healing process of the wart | After 1 treatment (Day 3 & Day 15), after 2 treatments (Day 30), after 3 treatments (Day 45)
  Evaluation of healing process of the wart by blinded dermatologist.
  This is done by assessing:
  * Discontinuation of skin lines (5 categories: 0=none, 1=light, 2=moderate, 3=severe, and 4=very severe)
  * Affection of skin color (5 categories: 0=none, 1=light, 2=moderate, 3=severe, and 4=very severe)
  * Presence/absence of a scab.
Local & general tolerance | When wart is considered cured at Day 15, Day 30 or Day 45 or at the end of study on Day 45.
  Evaluate the safety of the products by assessing local & general tolerance. Local tolerance will be assessed by using the following scale (0= Bad tolerance, 1= Moderade tolerance, 2= Good tolerance, 3=Very good tolerance.) Abnormal clinical signs and subjective signs reported by the subjects will be reported in the CRF.
  The general tolerance is a collection of adverse events by the investigator.

CONTACTS AND LOCATIONS:
Overall Officials: Ewa KARAMON, Principal Investigator — ewaczek20@wp.pl
Locations (1):
- Dermscan Poland, Gdansk, Poland